CLINICAL TRIAL: NCT00177268
Title: Peripheral Blood, Urine and Skin Sample Collection for Cutaneous Lymphoma, Eczema, and Atopic Dermatitis Research
Brief Title: Blood, Urine, and Tissue Collection for Cutaneous Lymphoma, Eczema, and Atopic Dermatitis Research
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Oleg E. Akilov, MD, PhD, Assistant Professor of Dermatology, University of Pittsburgh
Other Study IDs: STUDY19010322
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides; Eczema; Atopic Dermatitis
Keywords: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides; Blood/tissue banking; eczema; atopic dermatitis
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Mycosis Fungoides; Eczema; Dermatitis, Atopic | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — White blood cells and/or skin biopsy tissue are retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CTCL, atopic dermatitis, eczema: Those subjects with cutaneous t-cell lymphoma and Sezary syndrome, atopic dermatitis, or eczema may participate as appropriate with the potential for blood, tissue or urine sampling.
  Interventions: Other: Blood draw, skin biopsy or urine collection

INTERVENTIONS:
Other: Blood draw, skin biopsy or urine collection — Up to 9 blood draws/year of 60 ml of whole blood. One 6 mm punch biopsy may be obtained up to 4 times per year.

SUMMARY:
This is a tissue, urine, and blood banking protocol for cutaneous t-cell lymphoma (CTCL), eczema, and atopic dermatitis patients for current and future research.

DETAILED DESCRIPTION:
The purpose of this study is to provide a central mechanism for monitoring access to peripheral blood, urine, and skin specimens obtained from CTCL, eczema, and atopic dermatitis patients to monitor:

* immunologic assays/flow cytometry
* tumor progression/regression
* genomic studies
* proteomic studies
* others germane to the advancement of CTCL treatment

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* able and willing to provide informed consent
* diagnosed with CTCL
* diagnosed with either atopic dermatitis or eczema

Exclusion Criteria:

* Lack of CTCL, atopic dermatitis, or eczema diagnosis in medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with cutaneous t-cell lymphoma and/or Sezary syndrome and atopic dermatitis or eczema patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2004-10 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Proteomics of Cutaneous T-cell lymphoma | Ongoing
  Proteomic variables will be measured in blood and tissue of consented CTCL patients.

CONTACTS AND LOCATIONS:
Overall Officials: Oleg E Akilov, M.D., PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided